CLINICAL TRIAL: NCT01727687
Title: An Investigation of Road Crossing Safety Before and After Training Between Parkinson Disease Pedestrians and Older Pedestrians
Brief Title: Investigation of Road-crossing Safety Before and After Training Between Parkinson Disease Pedestrians and Older Pedestrians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PDcrossroad
Record Dates: First submitted 2012-01-02; First posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson's Disease
Keywords: To asses the training effects on traffic safety between normal and patients with Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Parkinson's disease (Experimental): Using simulated traffic scene system to help patients with Parkinson's disease improve crossing road behaviors.
  Interventions: Behavioral: behavioral training for crossing road

INTERVENTIONS:
Behavioral: behavioral training for crossing road — behavioral training programs for crossing road, such as verbal oral cues and simulated traffic scenes

SUMMARY:
As society ages, a large amount of human factors related research has been carried out into the subject of the safety of the elderly in their daily lives. However, most research focuses on the general elderly population and there is a serious lack of research into elderly sufferers of Parkinson's disease (PD), who receive a substantial amount of attention in medical circles. In the investigators previous study, the investigators have found that patient with PD had decreased ability to cross the road as compared to age/gender matched control subjects. Hence, this research proposed several training programs to enhance the safety of crossing road, including safe place finding，roadside search，time gap and perception of other's intentions. The investigators will compare the parameters of crossing road ability before and after training programs in patients with PD and control subjects.

The results of this research will clarify the correlation between medical scale test indicators and movement safety for patients with PD. The effects of training programs will be provided for further safety management and design concepts to improve the lives of this disease group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease
* Age between 18-80 years
* Patients signed the consent form

Exclusion Criteria:

* Patients with atypical parkinsonism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
The parameters of cross road | 1 year
  The main outcome variables were crossing time (CT), remaining time (RT), and safety margin (SM). The CT was the time taken by the subjects to cross the 3.5-m-wide road. The CT was measured at the normal walking pace and the fastest pace of each individual. Response time was measured in the simulated traffic situation and was defined as the time between starting the visual situation and the participant pressing the response button to decide to cross the road. The RT was the difference between the time gap (between the coming vehicle and the pedestrian) and the response time.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Hsien Lin, MD. PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan